CLINICAL TRIAL: NCT07268612
Title: A Phase 4 Retrospective Observational Study of CYFENDUS™ Anthrax Vaccine Among Individuals Who Received Post-Exposure Prophylaxis Vaccination During a Bacillus Anthracis Mass Exposure Event
Brief Title: Evaluation of Clinical Benefit and Safety Following CYFENDUS Administration for Post-Exposure Prophylaxis of Anthrax Disease.
Status: Not yet recruiting | Type: Observational
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Other Study IDs: EBS-AVA-213
Record Dates: First submitted 2025-11-24; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Anthrax
Keywords: Anthrax; Anthrax meningitis; cutaneous anthrax; gastrointestinal anthrax; inhalational anthrax; CYFENDUS; Anthrax vaccine adsorbed adjuvanted
MeSH Terms: conditions — Anthrax; Cutaneous anthrax; Gastrointestinal anthrax; Inhalation anthrax

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: CYFENDUS — Intramuscular administration of two doses of Anthrax Vaccine Adsorbed, Adjuvanted

SUMMARY:
The goal of this observational study is to evaluate the safety and clinical benefit of two doses of CYFENDUS vaccine when used with the concurrent recommended antibacterial regimen for post-exposure prophylaxis to prevent inhalational anthrax and/or anthrax meningitis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who received any dose of CYFENDUS vaccine (with or without concurrent recommended antibacterial regimen) for anthrax post exposure prophylaxis during an identified mass B. anthracis exposure event in the United States.

Exclusion Criteria:

* Individuals who did not receive CYFENDUS for anthrax post exposure prophylaxis during an identified mass B. anthracis exposure event in the United States.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include adults for which CYFENDUS is indicated (18 to 65 years of age), but it may include pediatric, pregnant, and geriatric populations if they are vaccinated with CYFENDUS based on public health recommendations as part of outbreak management.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2035-11 (Estimated); Primary Completion 2036-11 (Estimated); Study Completion 2037-11 (Estimated)

PRIMARY OUTCOMES:
Number of individuals who developed inhalational anthrax and/or anthrax meningitis and received CYFENDUS for post exposure prophylaxis divided by the total number reported to have received CYFENDUS for post exposure prophylaxis. | At least 12 months after containment of the mass exposure event